CLINICAL TRIAL: NCT02223377
Title: Most Effective Opioid Analgesia in Ambulatory Surgeries: a Randomized Control, Investigator Blinded, Parallel Group With Superiority Design Study of Morphine Versus Hydromorphone
Brief Title: Satisfactory Analgesia Minimal Emesis in Day Surgeries
Acronym: SAME-Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-482; CAS-2014-038 (Other Grant/Funding Number: AbbVie New Investigator's Award, CAS)
Record Dates: First submitted 2014-08-19; First posted 2014-08-22 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-03

CONDITIONS: Pain; Post Operative Nausea and Vomiting
MeSH Terms: conditions — Pain; Vomiting | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): Analgesia with equipotent doses of Morphine and Hydromorphone will be administered in titrated doses. Doses are 1ml=1mg of morphine or 0.2 mg of hydromorphone. Potency ratio of 1:5 (M: HM).
  0.05mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml)
  Interventions: Drug: Morphine
- Hydromorphone (Active Comparator): Analgesia with equipotent doses of Morphine and Hydromorphone will be administered in titrated doses. Doses are 1ml=1mg of morphine or 0.2 mg of hydromorphone. Potency ratio of 1:5 (M: HM).
  0.05mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml)
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Morphine — 1st dose: syringe of 0.04mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml); with a maximum of 3 mg of morphine equivalents is administered. Repeat doses: 0.02 mg/kg morphine units every 5-10 minutes to titrate for analgesia and side effects (rounding off to the nearest 1 ml or 0.5 ml)
  Other Names: Sandoz
  Arms: Morphine
Drug: Hydromorphone — 1st dose: syringe of 0.04mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml); with a maximum of 3 mg of morphine equivalents is administered. Repeat doses: 0.02 mg/kg morphine units every 5-10 minutes to titrate for analgesia and side effects (rounding off to the nearest 1 ml or 0.5 ml)
  Other Names: Sandoz
  Arms: Hydromorphone

SUMMARY:
Currently nearly 70% or more surgeries are being done as ambulatory (day care) procedures as they offer significant benefit to the patients as well as to the hospitals. Inadequate pain relief (30%-40%) and nausea-vomiting form the leading factors affecting the quality of care and hence its efficiency. Opioids form the primary modality to treat moderate to severe pain, but can also cause significant nausea-vomiting and other side effects. Although hydromorphone is five times more potent than morphine, in equianalgesic doses they both could provide similar pain relief. They both exert no ceiling effect for their analgesia, and hence incomplete or inadequate analgesia is related to the appearance of side effects. In this study the investigators shall assess the proportion of patients who satisfy the outcome of 'satisfactory analgesia with minimal nausea-vomiting' in ambulatory surgeries, assessed at 2 hours after surgery. Patients would be randomized to receive either morphine or hydromorphone in the surgical recovery area. All personnel involved with the study would be blinded. The investigators will also look to assess the time to discharge and other side effects. This will help to choose the better drug, thereby improving pain relief and side effects, and also the efficiency of health care delivery.

DETAILED DESCRIPTION:
There has been an exponential increase in the number of day case surgical procedures also called as ambulatory surgeries (AS), over the last 2 years.(1) Currently around 70% of procedures are being done as AS, with known benefits to patients and hospitals.(2) Its efficiency and cost effectiveness depends upon its organization and delivery of services. Pain and PONV are recognized as the leading factors affecting the quality of services delivered under AS,(1,3) and they affect the recovery, discharge, and overall satisfaction of patients.(4,5) According to literature, postsurgical pain could be inadequately treated in 30%-60% of patients and 30%-40% of AS patients suffer from significant PONV.(3,6,7) It is estimated that a single episode of PONV can prolong the PACU stay by 25 mins,(8) and patients rate PONV to be the most undesirable outcome associated with anesthesia.(4) Despite the increasing use of non-opioid analgesics, opioid analgesics have remained the primary modality in moderate to severe pain.(7) They cause several side effects such as drowsiness, sedation, PONV, itching and respiratory depression. Appropriate selection of opioid medications becomes significantly important to deliver safe and effective analgesia with minimal side effects. Although M has been the most commonly used medication, HM is also being increasingly used.(9) We do not yet know whether HM is more effective than M in AS patients. Both M and HM exert no ceiling effect for their analgesia, and by this nature incomplete or inadequate analgesia is related to the appearance of side effects.(10) Hence clinical effectiveness of opioids, relative to each other, is reflected not just by satisfactory analgesia, but by a combination of 'satisfactory analgesia with limited side effects'. Clinical observation suggests that HM is clinically better by providing superior or equivalent analgesia with decreased side effects.(9) HM is a semi-synthetic morphine derivative that differs from M in its position 6 of the benzol ring, where it has a keto-group instead of a hydroxy group, making it 5-10 times more potent and enhances its distribution to cerebral tissues, making for easier titration.(9) The t1/2 Ke0 (transfer life from plasma to effect site) is 1.6hr - 4 hr for M, compared to 18-38 min for HM.(9,10) It is observed that health care providers may be willing to provide higher dose of HM compared to M in EMU, as its actual quantity of drug is much smaller and therefore appears to cause less concern.(12, 13) Our literature review showed that there are no previous studies comparing these 2 medications in AS patients. The lone systematic review compared various acute and chronic pain studies, in various routes of drug administration.(9) Of the 11 studies identified; only 4 were done in acute pain settings.(13-16) Two of them were done by the same author in ER settings. Chang et al noted that HM reduced the mean pain scores by 1.3 units [95% CI= (-2.2 to -0.5)] compared to M in 198 adults treated in ER.(12,13). However it did not show much difference in geriatric population.14 In perioperative settings, Hong et al studied the difference in nausea between the 2 medications in 50 patients using PCA and found no difference.(15) Rapp et al studied various effects between the 2 medications in 61 surgical patients using PCA. There is not much clarity about their primary outcome; however they found the effects to be similar.(16) Both these studies had smaller sample sizes. The meta-analysis performed demonstrated that the HM does provide better analgesia than M, with a small effect size; Cohen's d=0.266 (p=0.012).(9) Looked at acute pain alone it was statistically significant (p=0.006), compared to chronic pain (p=0.889). It was noted that that there is a definite lack of comparative studies between them in surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory surgeries producing at least moderate pain-such as cholecystectomy, appendicectomy, ovarian cystectomy, inguinal hernia repair, abdominal wall hernias
* ability to communicate in English.

Exclusion Criteria:

* allergy to M or HM
* patient on regular chronic opioid medication
* patient uncontrolled systemic disease
* severe obesity with a BMI >35
* significant psychological impairment
* history of drug addiction or dependence
* any planned regional or nerve block other than local anesthesia infiltration patients with confirmed sleep apnea
* emergency surgeries and urological surgeries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2015-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Shanthanna, MD, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster University; James Paul, MD, Principal Investigator — Hamilton Health Sciences/McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario

REFERENCES:
- [Background] Sarin P, Philip BK, Mitani A, Eappen S, Urman RD. Specialized ambulatory anesthesia teams contribute to decreased ambulatory surgery recovery room length of stay. Ochsner J. 2012 Summer;12(2):94-100. PMID 22778673
- [Background] Troy AM, Cunningham AJ. Ambulatory surgery: an overview. Curr Opin Anaesthesiol. 2002 Dec;15(6):647-57. doi: 10.1097/00001503-200212000-00008. PMID 17019266
- [Background] Shnaider I, Chung F. Outcomes in day surgery. Curr Opin Anaesthesiol. 2006 Dec;19(6):622-9. doi: 10.1097/ACO.0b013e328010107e. PMID 17093366
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Background] Chatterjee S, Rudra A, Sengupta S. Current concepts in the management of postoperative nausea and vomiting. Anesthesiol Res Pract. 2011;2011:748031. doi: 10.1155/2011/748031. Epub 2011 Nov 3. PMID 22110499
- [Background] White PF. Pain management after ambulatory surgery - where is the disconnect? Can J Anaesth. 2008 Apr;55(4):201-7. doi: 10.1007/BF03021503. No abstract available. English, French. PMID 18378964
- [Background] Felden L, Walter C, Harder S, Treede RD, Kayser H, Drover D, Geisslinger G, Lotsch J. Comparative clinical effects of hydromorphone and morphine: a meta-analysis. Br J Anaesth. 2011 Sep;107(3):319-28. doi: 10.1093/bja/aer232. Epub 2011 Aug 5. PMID 21841049
- [Derived] Shanthanna H, Khaled MATM, Diaz A, Farsinejad P, Clements S. Low-dose remifentanil as an adjunct analgesic is not associated with clinically important opioid-induced hyperalgesia: secondary analysis from a randomized controlled trial. Reg Anesth Pain Med. 2025 Apr 24:rapm-2025-106483. doi: 10.1136/rapm-2025-106483. Online ahead of print. PMID 40274406
- [Derived] Shanthanna H, Paul J, Lovrics P, Vanniyasingam T, Devereaux PJ, Bhandari M, Thabane L. Satisfactory analgesia with minimal emesis in day surgeries: a randomised controlled trial of morphine versus hydromorphone. Br J Anaesth. 2019 Jun;122(6):e107-e113. doi: 10.1016/j.bja.2019.03.036. Epub 2019 Apr 23. PMID 31027915
- [Derived] Shanthanna H, Paul J, Lovrics P, Devereaux PJ, Bhandari M, Thabane L. Satisfactory Analgesia with Minimal Emesis in Day Surgeries (SAME DayS): a protocol for a randomised controlled trial of morphine versus hydromorphone. BMJ Open. 2018 Jun 22;8(6):e022504. doi: 10.1136/bmjopen-2018-022504. PMID 29934395

RESULTS

PARTICIPANT FLOW:
Groups:
- Morphine: Analgesia with equipotent doses of Morphine and Hydromorphone will be administered in titrated doses. Doses are 1ml=1mg of morphine or 0.2 mg of hydromorphone. Potency ratio of 1:5 (M: HM).
  0.05mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml)
  Morphine: Participant to be asked for their pain score, and if it is more than 4 out of 10 (NAS): to receive the 1st dose within 5 minutes after coming to PACU: 0.04mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml); with a maximum of 3 mg of morphine equivalents. Repeat doses: 0.02 mg/kg morphine units every 5-10 minutes to titrate for analgesia and side effects (rounding off to the nearest 1 ml or 0.5 ml)
- Hydromorphone: Analgesia with equipotent doses of Morphine and Hydromorphone will be administered in titrated doses. Doses are 1ml=1mg of morphine or 0.2 mg of hydromorphone. Potency ratio of 1:5 (M: HM).
  0.05mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml)
  Hydromorphone: Participant to be asked for their pain score, and if it is more than 4 out of 10 (NAS): to receive the 1st dose within 5 minutes after coming to PACU: 0.04mg/kg morphine units (rounding off to the nearest 1 ml or 0.5 ml); with a maximum of 3 mg of morphine equivalents. Repeat doses: 0.02 mg/kg morphine units every 5-10 minutes to titrate for analgesia and side effects (rounding off to the nearest 1 ml or 0.5 ml)
Period: Overall Study
Arm/Group | Morphine | Hydromorphone
Started | 199 | 203
Completed | 199 | 203
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Hydromorphone | Total
Number analyzed (Participants) | 199 | 203 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 175 | 357
  >=65 years | 17 | 28 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (13.8) | 47.1 (14.0) | 46.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 126 | 258
  Male | 67 | 77 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 199 | 203 | 402
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Patient's weight in kilograms (kg) divided by the square of patient's height in meters (m^2). (kg/m^2 ) Patients with BMI > 35 kg/m^2 are excluded from the study
  kg/m^2 | 27.55 (4.00) | 27.06 (4.27) | 27.37 (4.14)
Apfel score [Mean (Standard Deviation); unit: units on a scale] — The Apfel score is used as a predictor of postoperative nausea/vomiting (baseline variable).
  Four variables are scored as 0 or 1: 1) Postoperative opioids; 2) Non-smoker; 3) Female sex; 4) history of postoperative nausea/vomiting or motion sickness
  Scores range from 0 (10% risk of postoperative nausea/vomiting to 4 (80% risk of postoperative nausea/vomiting)
  When 0, 1, 2, 3, or 4 factors are present, the risk of PONV is 10%, 20%, 40%, 60%, or 80%, respectively
  units on a scale | 2.6 (0.9) | 2.5 (1.0) | 2.6 (0.9)
Depression score [Median (Inter-Quartile Range); unit: units on a scale] — Hospital Anxiety and Depression Scale. A 14-item measure (patient questionnaire) designed to assess anxiety and depression symptoms in medical patients.
  The Depression subscale has 7 statements with 4 possible responses each. Responses are scored from 0 (not at all) to 3 (always/very often/most of the time), with higher scores indicating worse depression. Max/min score for Depression subscale is 21/0.
  Scoring:
  Total score: Depression (D) ___________ 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
  units on a scale | 2 [1 to 5] | 2 [1 to 4] | 2 [1 to 4]
Anxiety score [Median (Inter-Quartile Range); unit: units on a scale] — Hospital Anxiety and Depression Scale. A 14-item measure (patient questionnaire) designed to assess anxiety and depression symptoms in medical patients.
  The Anxiety subscale has 7 statements with 4 possible responses each. Responses are scored from 0 (not at all) to 3 (always/very often/most of the time), with higher scores indicating worse anxiety. Max/min score for Anxiety subscale is 21/0.
  Scoring:
  Total score: Anxiety (A) ___________ 0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
  units on a scale | 6 [4 to 9] | 6 [3 to 8] | 6 [4 to 9]
Catastrophising score [Median (Inter-Quartile Range); unit: units on a scale] — Pain Catastrophizing Scale. This is a self-report measure, consisting of 13 items related to thoughts or feelings when experiencing pain, each item scored from 0 to 4 (0 - not at all; 1 - to a slight degree; 2 - to a moderate degree; 3 - to a great degree; 4 - all the time), resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
  units on a scale | 9 [1 to 17] | 10 [4 to 17] | 9 [3 to 17]
Preoperative pain in the operative area [Count of Participants; unit: Participants] — Presence of preoperative pain in the surgical area
  Participants | 83 | 83 | 166
Chronic pain in other areas [Count of Participants; unit: Participants] | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Our Combined Primary Outcome Will be Number of Patients With Same Analgesia Minimal Emesis, as Compared Between the 2 Groups.
Description: Our combined primary outcome will be number of patients with SAME, as compared between the 2 groups. Analgesia will be based on Numerical Analogue Scale for Pain 0-10 (appendix 3), and Post-operative nausea and vomiting will be based on Verbal Descriptive Scale 0-5 (appendix 3). These observations will be made at the end of 2 hrs or before (corresponding to the time of discharge from PACU), by the PACU nurse.
Time Frame: At 2hrs or at the time of discharge from PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 199 | 202
Participants | 172 | 175
Statistical Analysis 1: Comparison: Morphine vs Hydromorphone; Test type: Superiority; p = 0.997, Regression, Logistic; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.56 to 1.78]

2. Secondary Outcome: Number of Patients With Severe Itching
Description: Severe itching measured as visual analog scale score > 5 on a 0-10 Visual Analog Scale, where 0 = no itching, and 10 = worst itching imaginable
Time Frame: At 2hrs or at the time of discharge from PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 199 | 202
Participants | 2 | 5

3. Secondary Outcome: Severe Sedation
Description: Ramsay Sedation Scale 0-6
Time Frame: At 2hrs or at the time of discharge from PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 199 | 202
Participants | 5 | 8

4. Secondary Outcome: Severe Respiratory Depression
Description: Presence of Respiratory Rate below 10 and/or Presence of Oxygen Saturation <90
Time Frame: At 2hrs or at the time of discharge from PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 199 | 202
Participants | 11 | 10

5. Secondary Outcome: Patients Requesting Oral Analgesia in the Day Surgery Unit
Description: Use of rescue drug for pain
Time Frame: At 2hrs or at the time of discharge from PACU
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 194 | 199
Participants | 128 | 135

6. Secondary Outcome: Mean Dose of Analgesic Used
Description: For a day surgery case, from the time of hospital admittance to discharge from hospital is an average 5 hours.
Time Frame: 5 hours post-admit to hospital
Measure: Mean (Standard Deviation); unit: Equivalent morphine unit
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 199 | 202
Equivalent morphine unit | 5.7 (3.9) | 4.9 (3.3)
Statistical Analysis 1: Comparison: Morphine vs Hydromorphone; Test type: Superiority; p = 0.040, ANOVA; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.43 to -0.03]

7. Secondary Outcome: Patient Satisfaction Score
Description: Patient satisfaction is measured on a 0-10 visual analogue scale, where 0=completely unsatisfied; 10=extremely satisfied
Time Frame: At 5 hours post-admit to hospital
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 184 | 177
score on a scale | 9.1 (1.8) | 9.3 (1.2)

8. Secondary Outcome: Time to Discharge From PACU
Description: For a day surgery case, from the time out of operating room to discharge from PACU is an average 2 hours.
Time Frame: At 2hrs or at the time of discharge from PACU
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 198 | 201
Minutes | 91.2 (58.6) | 92.8 (50.6)

9. Secondary Outcome: Time to Discharge From Hospital
Description: For a day surgery case, from the time of hospital admittance to discharge from hospital is an average 5 hours.
Time Frame: At 5 hours post-admit to hospital
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Morphine | Hydromorphone
Number analyzed (Participants) | 199 | 197
Hours | 3.2 (1.1) | 3.3 (1.1)

ADVERSE EVENTS:
Time Frame: At 2 hours or at the time of discharge from PACU, and at 24 h after surgery
Arm/Group | Morphine | Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/202
Serious Adverse Events (participants affected / at risk) | 11/199 | 10/202
Other Adverse Events (participants affected / at risk) | 7/199 | 13/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (N=199) | Hydromorphone (N=202)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 11 | 10 — Proportion of patients with respiratory depression: patients needing naloxone treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Morphine (N=199) | Hydromorphone (N=202)
Severe itching (Skin and subcutaneous tissue disorders) | 2 | 5 — measured as visual analogue scale (VAS)>5/10.
Severe sedation (Nervous system disorders) | 5 | 8 — Proportion of patients with severe sedation: measured as Ramsay sedation score >3/6.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02223377/Prot_SAP_000.pdf